CLINICAL TRIAL: NCT06540339
Title: SnapPelvis: International Prospective Observational Cohort Study of Traumatic Pelvic Ring Injuries
Brief Title: A Snapshot Audit of Traumatic Pelvic Ring Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Aachen (Other)
Collaborators: European Society for Trauma and Emergency Surgery (Other)
Responsible Party: Principal Investigator, Dr. med. Eftychios Bolierakis, Dr. med. Eftychios Bolierakis, University Hospital, Aachen
Other Study IDs: 520741
Record Dates: First submitted 2024-07-20; First posted 2024-08-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Trauma; Pelvic Fracture; Fragility Fractures of the Pelvis (FFP)
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with high-energy pelvic ring injuries
  Interventions: Other: Snapshot-audit studies do not necessitate any intervention in the defined cohorts.
- Patients with complex pelvic trauma
  Interventions: Other: Snapshot-audit studies do not necessitate any intervention in the defined cohorts.
- Pratients with fragility fractures of the pelvis
  Interventions: Other: Snapshot-audit studies do not necessitate any intervention in the defined cohorts.

INTERVENTIONS:
Other: Snapshot-audit studies do not necessitate any intervention in the defined cohorts. — Snapshot-audit studies do not necessitate any intervention in the defined cohorts.

SUMMARY:
Multicenter, snapshot cohort studies or audits have the ability to gather large patient numbers in short time periods from many healthcare systems with different resources or practices of care concerning one specific surgical condition. This type of studies allows exploration of differences in patient populations and management across the sampled cohort to identify areas of practice variability that may result in apparent differences in outcome. As such, whilst not providing true evidence of efficacy or the impact of a single variable on overall outcome, these studies can be hypothesis-generating and identify areas warranting further study in future randomized controlled trials (1). Snapshots also shed light on the real world practice, rather than the presumed or guideline suggested patient care (2).

Traumatic Pelvic Ring Injuries (TPRI) represent a broad spectrum of trauma-associated pathologies with a distinct bimodal age distribution in patients admitted through the Emergency Departments of all acute care hospitals. In younger patients, this type of injury is often associated with high-energy trauma, hemodynamic instability, high mortality and morbidity rates (3-6). In the elderly population, pelvic fractures result from low energy trauma mechanisms (e.g. ground level fall) and can affect the long-term independency and life quality of geriatric patients (7).

There is substantial variation in the management of pelvic ring injuries among pelvic trauma surgeons; these variations include but are not limited to the timing of definitive fixation, the indications and protocols of conservative treatment, and the appropriate osteosynthesis of the anterior and/or posterior pelvic fractures (8).

This 'ESTES snapshot audit' -a prospective observational cohort study- has a dual purpose. Firstly, as an epidemiological study, it aims to report the burden of injury in specific hospitals, distributed widely throughout Europe. Secondly, this study aims to demonstrate current strategies for both, younger (after high-energy trauma) and geriatric patients (after low-energy trauma) employed to assess and treat these patients. These twin aims will serve to provide a 'snapshot' of current medical practice, but will also be hypothesis-generating while providing a rich source of patient-level data to allow further analysis of particular clinical questions. The acquired study data can be subsequently evaluated and compared to patient data of established pelvic trauma registries across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) admitted for traumatic pelvic ring injuries (AO/FFP-Classification).

Exclusion Criteria:

* Concomitant acetabular fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients diagnosed in the emergency department of participating hospitals across Europe with traumatic pelvic ring injuries over a 3-month period.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Mortality after traumatic pelvic ring injuries | 6 months

SECONDARY OUTCOMES:
Rate of systemic complications after traumatic pelvic ring injuries | 6 months
Re-admission rate for fracture-related implant failure, infections and re-operations within 6 months after traumatic pelvic ring injuries | 6 months
Pelvic Outcome Score after traumatic pelvic ring injuries | 6 months
  The Pelvic Outcome Score reflects the outcome after treatment of traumatic pelvic ring injuries. It assesses following three parameters: radiological result (max. 3 points), clinical result (max. 4 points) and social reintegration (max. 3 points). The maximum of 10 points represents an excellent result, while the minimum of 3 points corresponds to the worst outcome (9).
Rate of social reintegration after traumatic pelvic ring injuries | 6 months
  Rate of retaining same profession, recreational status, activity level in sports and social situation as prior to accident. This outcome measure will be assessed through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hildebrand, Prof. Dr., Study Chair — University Hospital, Aachen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bass GA, Kaplan LJ, Ryan EJ, Cao Y, Lane-Fall M, Duffy CC, Vail EA, Mohseni S. The snapshot audit methodology: design, implementation and analysis of prospective observational cohort studies in surgery. Eur J Trauma Emerg Surg. 2023 Feb;49(1):5-15. doi: 10.1007/s00068-022-02045-3. Epub 2022 Jul 15. PMID 35840703
- [Background] Bass GA, Gillis A, Cao Y, Mohseni S; European Society for Trauma, Emergency Surgery (ESTES) Cohort Studies Group. Patterns of prevalence and contemporary clinical management strategies in complicated acute biliary calculous disease: an ESTES 'snapshot audit' of practice. Eur J Trauma Emerg Surg. 2022 Feb;48(1):23-35. doi: 10.1007/s00068-020-01433-x. Epub 2020 Jul 7. PMID 32632631
- [Background] Enninghorst N, Toth L, King KL, McDougall D, Mackenzie S, Balogh ZJ. Acute definitive internal fixation of pelvic ring fractures in polytrauma patients: a feasible option. J Trauma. 2010 Apr;68(4):935-41. doi: 10.1097/TA.0b013e3181d27b48. PMID 20386287
- [Background] Ertel W, Keel M, Eid K, Platz A, Trentz O. Control of severe hemorrhage using C-clamp and pelvic packing in multiply injured patients with pelvic ring disruption. J Orthop Trauma. 2001 Sep-Oct;15(7):468-74. doi: 10.1097/00005131-200109000-00002. PMID 11602828
- [Background] Logters T, Lefering R, Schneppendahl J, Alldinger I, Witte I, Windolf J, Flohe S; TraumaRegister der DGU. [Interruption of the diagnostic algorithm and immediate surgical intervention after major trauma--incidence and clinical relevance. Analysis of the Trauma Register of the German Society for Trauma Surgery]. Unfallchirurg. 2010 Oct;113(10):832-8. doi: 10.1007/s00113-010-1772-1. German. PMID 20393832
- [Background] Timmer RA, Mostert CQB, Krijnen P, Meylaerts SAG, Schipper IB. The relation between surgical approaches for pelvic ring and acetabular fractures and postoperative complications: a systematic review. Eur J Trauma Emerg Surg. 2023 Apr;49(2):709-722. doi: 10.1007/s00068-022-02118-3. Epub 2022 Nov 25. PMID 36434301
- [Background] Kuper MA, Trulson A, Stuby FM, Stockle U. Pelvic ring fractures in the elderly. EFORT Open Rev. 2019 Jun 3;4(6):313-320. doi: 10.1302/2058-5241.4.180062. eCollection 2019 Jun. PMID 31312519
- [Background] Parry JA, Funk A, Heare A, Stacey S, Mauffrey C, Starr A, Crist B, Krettek C, Jones CB, Kleweno CP, Firoozabadi R, Sagi HC, Archdeacon M, Eastman J, Langford J, Oransky M, Martin M, Cole P, Giannoudis P, Byun SE, Morgan SJ, Smith W, Giordano V, Trikha V. An international survey of pelvic trauma surgeons on the management of pelvic ring injuries. Injury. 2021 Oct;52(10):2685-2692. doi: 10.1016/j.injury.2020.07.027. Epub 2020 Jul 11. PMID 32943214
- [Background] Pohlemann T, Gansslen A, Schellwald O, Culemann U, Tscherne H. Outcome after pelvic ring injuries. Injury. 1996;27 Suppl 2:B31-8. PMID 8915200